CLINICAL TRIAL: NCT00529490
Title: The Efficacy and Safety of Hypertonic Lactate Solution as Fluid Resuscitation Compared With Ringer's Lactate in Post-CABG (Coronary Artery Bypass Grafting) Patients
Brief Title: Efficacy, Safety of Hypertonic Lactate Soln. as Fluid Resuscitation Compared With Ringer's Lactate in Post-CABG Pats
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innogene Kalbiotech Pte. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001/CT-KB/DNA/02
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2007-09

CONDITIONS: Low Cardiac Output
Keywords: coronary; artery; bypass; grafting; I.V.; cardiac output
MeSH Terms: conditions — Cardiac Output, Low | interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HL (Experimental): Hypertonic lactate group
  Interventions: Drug: Hypertonic lactate
- RL (Active Comparator): Ringer's lactate
  Interventions: Drug: Ringer's lactate

INTERVENTIONS:
Drug: Hypertonic lactate — Parenteral solution administered to a maximal volume of 10 ml/kg BW over the first 12 hours post-CABG
  Other Names: Totilac
  Arms: HL
Drug: Ringer's lactate — Parenteral solution administered to a maximal dose of 30 ml/kg BW over the first 12 hours post-CABG
  Arms: RL

SUMMARY:
Prospective, randomized, open-label study to assess the efficacy and safety of hypertonic lactate solution, compared to Ringer's Lactate as fluid resuscitation to maintain hemodynamic stability in post-coronary artery bypass grafting(CABG) patients. Patients who were eligible received either hypertonic lactate solution or Ringer's Lactate post-CABG in the ICU when fluid resuscitation was needed.

DETAILED DESCRIPTION:
Prospective, randomized, open-label study to assess the efficacy and safety of hypertonic lactate solution, compared to Ringer's Lactate as fluid resuscitation to maintain hemodynamic stability in post-coronary artery bypass grafting(CABG) patients. Patients who were eligible received either hypertonic lactate solution or Ringer's Lactate post-CABG observed in the first 12 hours in the ICU when fluid resuscitation was needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given their written informed consent.
* Male or female, aged 18-75 years.
* Post-operative CABG on pump or off pump in ICU.
* Patients who need fluid resuscitation.

Exclusion Criteria:

* Combined operations.
* Need for intra aortic balloon pump (IABP).
* Patients with severe arrhythmia (VT, AF rapid response, heart block).
* Severe hemodynamic imbalance.
* Severe bleeding and/or re-operation.
* Liver dysfunction(SGOT and SGPT 2x normal).
* Renal failure (Creatinine >2 mg%).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2002-03; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
hemodynamic stability | 12 hours post-CABG surgery

SECONDARY OUTCOMES:
Safety of hypertonic sodium lactate for maintaining the hemodynamic stability | 12 hours post-CABG surgery

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Mustafa, MD, Principal Investigator — National cardiac Centre, Harapan Kita Hospital, Dept. of Anaesthesiology, Intensive Care Unit, Jakarta, Indonesia; Xavier Leverve, MD, PhD, Principal Investigator — Director, INSERM-E0221-Bioenergetique Fondamentale et Appliquée Université, Joseph Fourier, France
Locations (1):
- National Cardiac Center, Department of Surgery and Intensive Care Unit, Harapan Kita Hospital, Jakarta, Jakarta Special Capital Region, Indonesia